CLINICAL TRIAL: NCT05473104
Title: Program for the Education and Enrichment of Relational Skills (PEERS®) for Italy. A RCT's Study on Social Skills Intervention for Adolescents With Autism Spectrum Disorder (ASD).
Brief Title: PEERS® for Italy, a Study on Social Skills Intervention for Adolescents With Autism Spectrum Disorder (ASD).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Superiore di Sanità (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Laura Maria Fatta, Ph.D Psy.D, Istituto Superiore di Sanità
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 871
Record Dates: First submitted 2022-07-04; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; social skills training
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Teens and parents participate in the training once a week for 14 consecutive weeks in parallel groups.
  Interventions: Behavioral: Program for the Education and Enrichment of Relational Skills
- waiting-list group (No Intervention): Teens and parents participate in the training in a second moment, immediately after the experimental group concluded the program, once a week for 14 consecutive weeks in parallel groups.

INTERVENTIONS:
Behavioral: Program for the Education and Enrichment of Relational Skills — Social training targeting adolescents with ASD and focused on making and keeping friends
  Arms: experimental group

SUMMARY:
TThe research aims to verify the Italian adaptation of a parent-mediated group training focused on social skills for adolescents with autism spectrum disorder (ASD). The Program for the Education and Enrichment of Relational Skills PEERS® is an evidence-based program with substantial literature (over 40 studies) applied in several countries. For the present study, about 40 adolescents, both boys, and girls with ASD, are enrolled and randomized into two groups. Groups (experimental group and waiting list) took part in the Italian telehealth adaptation of PEERS® at different times and were evaluated at several time points (baseline, pre-treatment, post-treatment, and follow-up). The objective of the comparison was to explore the primary outcomes, such as the impact of training on social knowledge and performance, and secondary outcomes, like psychiatric comorbidities and neuropsychological profile. The hypothesis is that social skills (knowledge and performance) improve after training in the experimental group and affect the secondary outcomes, and the achievements are maintained at 3-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* a previous and current diagnosis of ASD, by a clinical team, according to DSM-5, clinical observation and structured assessment with standardized tests (Autism Diagnostic Observation Schedule- Second Edition; ADOS-2; Lord et al., 2012)
* Verbal Comprehension Index scores at least 80 on the Italian version of the WISC-IV scale (Orsini et al.,2012).
* Chronological age between 12 and 18 years;
* Social problems as reported both by the parents and adolescents;
* Italian fluency for the adolescent and parent
* Abstention from other social skills training (following a manualized protocol).
* No history of adolescent major mental illness, such as bipolar disorder, schizophrenia, or psychosis;
* No history of hearing, visual, or physical impairmentsExclusion Criteria:

Exclusion Criteria:

* No diagnosis of ASD.
* IQ Total score below 70 or Verbal Comprehension Index scores below 80 on the Italian version of the WISC-IV scale (Orsini et al.,2012).
* Lack of motivation (both parents or adolescents).
* Participation in another social skills training (following a manualized protocol).
* Auto-aggressive behaviors

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Social Responsiveness Scale (SRS) (Costantino & Gruber, 2005), changes after 14 weeks and 3 months. | pre-treatment, after 14 weeks and 3 months after the start of training (within two weeks)
  is a quantitative measure completed by caregivers and teachers, consisting of 65 items, assessing symptoms characteristic of autism spectrum disorders, in children and adolescents aged 4 to 18 years. In this study it is used as a primary outcome measure to assess global social skills.
Quality of Socialization Questionnaire-Revised (QSQ-R) (Laugeson & Frankel, 2010; Laugeson et al., 2012), changes after 14 weeks and 3 months. | pre-treatment, after 14 weeks and 3 months after the start of training (within two weeks)
  It is a social performance measure filled out both by caregivers and adolescents, assessing, through numbers and quality of get-togethers, the ability to know how to make and maintain friendships in the natural contexts of adolescents.
Test of Adolescent Social Skills Knowledge (TASSK) (Laugeson & Frankel 2010), changes after 14 weeks and 3 months. | pre-treatment, after 14 weeks and 3 months after the start of training (within two weeks)
  It is a 30-question questionnaire completed by adolescents to monitor the acquisition of the topics covered within the PEERS®. It is used to evaluate social knowledge.assessing, through numbers and quality of get-togethers, the ability to know how to make and maintain friendships in the natural contexts of adolescents.

SECONDARY OUTCOMES:
Child Behavior Checklist (CBCL) (Achenbach & Rescorla, 2001), changes after 14 weeks and 3 months. | pre-treatment, after 14 weeks and 3 months after the start of training (within two weeks)
  CBCL is widely used to evaluate developmental psychopathology through scales that assess specific dimensions (Anxiety/Depression; Withdrawal/Depression; Somatic Complaints; Social Problems; Thinking Problems; Attention Problems; Rule-Breaking Behaviors; Aggressive Behaviors), general (Internalizing, Externalizing, and Total Problems), emotional-behavioral problems according to some of the DSM diagnostic categories (Affective Problems; Anxiety Problems; Somatic Problems; Attention-Deficit/Hyperactivity Problems; Oppositional-Provocative Problems; Conduct Problems). We used parent, teacher, and adolescent forms
Multidimensional Anxiety Scale for Children-Second Edition (MASC-2) (March, 2013), changes after 14 weeks and 3 months. | pre-treatment, after 14 weeks and 3 months after the start of training (within two weeks)
  It is a 50-item questionnaire completed by adolescents, assessing anxiety in children and adolescents from 8 to 19 years of age comprehensively.
Children's Depression Inventory, Second Edition (CDI-2) (Kovacs, 2010), changes after 14 weeks and 3 months. | pre-treatment, after 14 weeks and 3 months after the start of training (within two weeks)
  It is a comprehensive, multi-perspective assessment of depressive symptoms in children and adolescents aged 7 to 17 years that allows early identification of depressive symptoms and provides an index of their extent and severity. We used the children and adolescent version
Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) (Gioia et al., 2015), changes after 14 weeks and 3 months. | pre-treatment, after 14 weeks and 3 months after the start of training (within two weeks)
  ICompleted by caregivers, assessing the executive functioning profile of children between the ages of 5 and 18 years oldand adolescents aged 7 to 17 years that allows early identification of depressive symptoms and provides an index of their extent and severity. We used the children and adolescent version

OTHER OUTCOMES:
Autism Quotient (AQ) (Baron-Cohen et al., 2001) | pre-treatment (within two weeks)
  It was administered to parents separately to evaluate autism traits.
Adaptive Behavior Assessment System - Second Edition (ABAS-II) (Harrison & Oakland 2003) | pre-treatment (within two weeks)
  It is a rating scale that measures daily living skills. It can detect these skills in individuals aged 0-89 years. For the present study, the caregivers' form was used to assess the behavior of people aged 5 to 21.
Social validity | post-treatment (within two weeks)
  The questionnaire was administered to adolescents, and caregivers to evaluate the usefulness of the program sessions (using a 3-point likert scale) and whether they would recommend the training to other families/peers. Finally, they were asked to indicate 3 strengths and 3 weaknesses. The questionnaires were constructed specifically for the current research project from a reworking of a form found in another study that used PEERS® to test the program's effectiveness with participants with Turner Syndrome (Wolstencroft et al., 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Superiore di Sanità, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fatta LM, Laugeson EA, Bianchi D; Italian Peers(R) team support group; Laghi F, Scattoni ML. Program for the Education and Enrichment of Relational Skills (PEERS(R)) for Italy: A Randomized Controlled Trial of a Social Skills Intervention for Autistic Adolescents. J Autism Dev Disord. 2025 Jan;55(1):202-220. doi: 10.1007/s10803-023-06211-3. Epub 2024 Jan 8. PMID 38190054